CLINICAL TRIAL: NCT06938334
Title: A Single-arm, Open-label, Phase I/II Clinical Trial of Autologous Hematopoietic Stem and Progenitor Cells (HSPCs) Genetically Modified With a Lentiviral Vector (LVV) Encoding for the Human Programmed Death-ligand 1 (hPD-L1) Complementary Deoxyribonucleic Acid (cDNA) for the Treatment of Patients With Type 1 Diabetes (T1D) at Recent Onset and With Residual β-cell Function (IMMUNOSTEM)
Brief Title: A First-in-human Clinical Trial Using a Gene Therapy With Patient's Own Stem Cells to Treat Early Type 1 Diabetes
Acronym: IMMUNOSTEM
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Altheia Science (Industry)
Collaborators: Evidenze Health S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMUNOSTEM; 2025-521304-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Diabetes, Type I
Keywords: type 1 diabetes (T1D); HSPCs genetically modified; lentiviral vector (LVV)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Evaluation of the safety and efficacy of autologous CD34+ HSPCs transduced ex vivo with LVV encoding hPD-L1 cDNA in patients with T1D at recent onset and with residual β-cell function
  Interventions: Genetic: Autologous CD34+ cell enriched population containing HSPCs transduced ex vivo using a LVV encoding the hPD-L1 DNA

INTERVENTIONS:
Genetic: Autologous CD34+ cell enriched population containing HSPCs transduced ex vivo using a LVV encoding the hPD-L1 DNA — The intervention is intended for newly diagnosed T1D patients with residual beta-cell function, who can receive the Drug Product (DP) within 180 days from the first insulin administration. Mobilized autologous HSPCs, collected by leukapheresis, are ex vivo transduced with a LVV encoding for hPD-L1 and formulated in a cryopreservation medium containing DMSO (DP). After release, the DP is thawed and administered to the patient at a dose ranging between 5 and 20 million of cells per kilogram of body weight. The intervention plans for a single DP injection.

SUMMARY:
Purpose:

The purpose of the trial is to assess the safety profile of the study treatment and to evaluate its efficacy in terms of improvement in key diabetes management parameters, including insulin requirements and β-cell function, and immunological parameters, in patients with T1D at recent onset / diagnosis and with residual β-cell function.

Rationale:

The study treatment consists of an autologous CD34+-enriched population that contains HSPCs transduced ex vivo with a third generation VSV-G pseudotyped LVV encoding the hPD-L1 cDNA. The drug product (DP) is composed of genetically modified autologous CD34+ HSPCs formulated in cryopreservation medium, transferred to the final container closure, and cryopreserved.

The mechanism of action is based on the ability of the PD-L1-expressing HSPCs to exert immunoregulatory properties activity and ablate suppress the autoimmune reaction induced by auto-reactive T lymphocytes, by homing to the site of inflammation, i.e., the pancreas.

PD-L1 is the ligand for the PD-1 receptor, expressed primarily on activated T cells. Crosslinking of PD-L1 and PD-1 inhibits T cell activation and favours their exhaustion/apoptosis and in mice deficient in PD-L1/PD-1 develop accelerated diabetes. HSPCs have been extensively used as an effective therapeutic approach in haematological malignancies and have demonstrated to be safe in human subjects.

Immunologically based clinical trials performed thus far have failed to cure T1D, in part because these approaches were nonspecific. Because the disease is driven by autoreactive CD4+ T cells, which destroy β cells, transplantation of hematopoietic stem and progenitor cells (HSPCs) has been recently offered as a therapy for T1D. Our transcriptomic profiling of HSPCs revealed that these cells are deficient in PD-L1, an important immune checkpoint, in the T1D non-obese diabetic (NOD) mouse model. Notably, the immunoregulatory molecule PD-L1 plays a determinant role in controlling/inhibiting activated T cells and thus maintains immune tolerance. Furthermore, our genome-wide and bioinformatic analysis revealed the existence of a network of microRNAs (miRNAs) controlling PD-L1 expression, and silencing one of key altered miRNAs restored PD-L1 expression in HSPCs. The Investigators therefore sought to determine whether restoration of this defect would cure T1D as an alternative to immunosuppression. Genetically engineered or pharmacologically modulated HSPCs overexpressing PD-L1 inhibited the autoimmune response in vitro, reverted diabetes in newly hyperglycemic NOD mice in vivo, and homed to the pancreas of hyperglycemic NOD mice. The PD-L1 expression defect was confirmed in human HSPCs in T1D patients as well, and pharmacologically modulated human HSPCs also inhibited the autoimmune response in vitro.

The Investigators therefore hypothesized that targeting a specific immune checkpoint defect in HSPCs thus may contribute to establishing a cure for T1D or slow the progression of β-cell destruction.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, compliance with the requirements and restrictions listed in the Informed Consent Form and the protocol.
2. Male and or female patients.
3. Age ≥18 and ≤40 years
4. Patient able to comply with all protocol procedures for the duration of the study.
5. Recent T1D onset/diagnosis (patients should receive the DP within 180 days from the 1st insulin administration).
6. HbA1c ≥53 and ≤150 mmol/mol
7. Positivity to at least 2 autoantibodies (i.e., anti-insulin, IAA; anti-glutamic acid decarboxylase 65, GAD65; anti-islet antigen 2, IA-2A; anti-zinc transporter 8, ZnT8; anti-islet cell antibody, ICA).
8. Basal C-peptide levels ≥0.2 nmol/L or ≥0.6 ng/mL; if basal C-peptide levels <0.2 nmol/L, stimulated C-peptide peak ≥0.2 nmol/L or ≥0.6 ng/mL during a 2-hour MMTT; MMTT should not be performed within one week of resolution of a diabetic ketoacidosis event.

Exclusion Criteria:

1. Unwillingness to sign the informed consent.
2. Type 2 diabetes
3. Any other unstable chronic disease
4. Significant systemic infection during the four weeks before requiring hospitalisation, administration of intravenous antibiotics, surgery
5. Present administration of chemotherapeutic anti-neoplastic drugs.
6. QTcF >470 msec.
7. Occurrence of an episode of ketoacidosis or hypoglycaemic coma in the past two weeks.
8. Presence of a ≥grade 3 adverse event (including laboratory analyses) according to CTCAE version 5.0.
9. Evidence of clinically significant abnormalities at bone-marrow aspirate
10. Body Mass Index (body weight*height2 )>27 kg⁄m2
11. A positive result to Biological Screening testing for Anti-HCV Antibody (Ab), HCV nucleic acid test (NAT) (if anti-HCV Ab positive), HIV-1/-2 p24 Ab and antigen (Ag), HIV RNA NAT, anti-Treponema pallidum total Ig, HbsAg (Australia Ag), HBV DNA NAT, total anti-HB core Ab (if HBV DNA NAT positive), anti-HTLV I, and anti-HTLV II (if applicable).
12. Active SARS-CoV-2 infection.
13. Allergy to mobilizing agents (G-CSF and plerixafor).
14. Pregnancy or lactation
15. Absence of an efficacious method of contraception
16. Any condition that in the opinion of investigator contraindicate apheresis or infusion of transduced HSPCs or affects patient's compliance.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Up to 24 months
  For each participant, number, description and grading of any adverse event, including expected and unexpected adverse events, meeting or not meeting the definition of "serious".

SECONDARY OUTCOMES:
Vector Copy Number | Up to 24 months
  Longitudinal analysis of vector copy number (VCN) in peripheral blood samples to assess frequency and persistence of infused cells and their progenies
Safety and efficacy | on month 12 and 24 month
  Changes over time of the 3-hour area under curve (AUC) and ΔAUC normalised by baseline glucose blood levels of C-peptide response to a mixed meal tolerance test (MMTT) over 12 and 24 months
Safety and efficacy | on month 12 and 24 month
  Changes over time of glucose metrics from continuous glucose monitoring (CGM) over 12 and 24 months
Safety and efficacy | Up to 24 months
  Exogenous insulin requirement defined as a daily average in units per kilogram per day (U/kg/day) during the previous 14 days
Pharmacodynamic | from Treatment to end of study
  Longitudinal analysis of vector copy number (VCN) in peripheral blood samples to assess frequency and persistence of infused cells and their progenies
Safety and efficacy | on month 12 and 24 month
  Changes over time of HbA1c levels over 12 and 24 months
Safety and efficacy | Up to 24 months
  Number of self-reported episodes of severe (CTCAE version 5.0 grade 3) hypoglycaemia

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale-Università Padova, Padua, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: June 2029 - June 2030

REFERENCES:
- [Background] Ben Nasr M, Tezza S, D'Addio F, Mameli C, Usuelli V, Maestroni A, Corradi D, Belletti S, Albarello L, Becchi G, Fadini GP, Schuetz C, Markmann J, Wasserfall C, Zon L, Zuccotti GV, Fiorina P. PD-L1 genetic overexpression or pharmacological restoration in hematopoietic stem and progenitor cells reverses autoimmune diabetes. Sci Transl Med. 2017 Nov 15;9(416):eaam7543. doi: 10.1126/scitranslmed.aam7543. PMID 29141886